CLINICAL TRIAL: NCT01531608
Title: Evaluation Of Mobile Gamma Camera Imaging For Sentinel Node Biopsy In Melanoma Independent Of Fixed Gamma Camera Imaging
Brief Title: Evaluation Of Mobile Gamma Camera Imaging For Sentinel Node Biopsy In Melanoma
Acronym: Mel54
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Craig L Slingluff, Jr, Professor, Department of Surgery, University of Virginia
Other Study IDs: 15343
Record Dates: First submitted 2012-01-30; First posted 2012-02-13 (Estimated); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Melanoma
Keywords: melanoma; imaging; sentinel node; biopsy
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a single-institution study seeking to evaluate if mobile gamma camera imaging can be used independent of standard fixed gamma camera imaging in patients undergoing sentinel node biopsy for melanoma.

DETAILED DESCRIPTION:
Patients who are scheduled to undergo sentinel node biopsy as part of recommended clinical care will be offered participation in this study.

Patients enrolled in this study will receive standard lymphoscintigraphy in nuclear medicine; however, these images will not be reviewed by the investigator until the preoperative mobile gamma camera(MGC)images have been obtained. Upon completion of the preoperative MGC imaging, the investigator will define the location of SLNs and the plan for the surgical approach. The investigator will then review the FGC images and assess the agreement of these two imaging methodologies. The hand-held gamma probe will be used to further evaluate the patient at this time and a final determination of true hot spots will be made based on the information and the clinical judgment of the operating surgeon. The final surgical plan will be decided. The primary data to be obtained from this cohort will be confirmation of the use of MGC imaging as a screening device to identify all nodal basins containing SLNs.

An additional goal of this study will be to identify techniques that may improve the use of the MGC and opportunities for optimizing the MGC device and imaging system. To the extent possible, improvements to the system will be made incrementally. A goal is to have a more optimized system before the next trial.

In addition to the preoperative imaging data discussed above, the participants will be reevaluated intraoperatively with a MGC and the hand-held probe at the following time points:

1. after removal of each sentinel node
2. after completion of the sentinel node biopsy procedure In each of these assessments, the following will be recorded: the number and location of sentinel nodes, the correspondence with preoperative hot spots determined by the clinical gamma detection devices (fixed camera, MGC and hand-held probe), the time required for imaging, and technical features of use, advantages, and limitations of the MGC imaging system. The individual sentinel nodes will be imaged ex vivo and counted with the hand-held probe.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of melanoma for whom a sentinel node biopsy is planned as part of standard surgical management of the melanoma. Patients may have more than one primary lesion.
* Patients with other malignancies may be included in this study, but the primary focus of this study is on melanoma, and data analysis of the melanoma patients will be independent of patients for whom sentinel node biopsy is done for other malignancies. It may also include patients for whom the diagnosis of melanoma is not certain but sentinel node biopsy is planned as part of the standard management (e.g.: severely atypical melanocytic neoplasms of uncertain malignant potential).
* All patients must have the ability and willingness to give informed consent.
* Age 18 years or older at the time of study entry. (Younger patients are excluded for simplicity since this avoids the requirement for separate consent documents, this is just a pilot study, and patients under age 18 are uncommon enough that they would not be likely to be enrolled in this small pilot study)

Exclusion Criteria:

* Participants in whom there is a medical contraindication or potential problem in complying with the requirements of the protocol in the opinion of the investigator
* Patients receiving there technetium injection more than 12 hours prior to their scheduled surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with melanoma scheduled to undergo sentinel node biopsy as part of recommended clinical care, age 18 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-03; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Identification of "misses" in which the operative approach was altered using data from the FGC. | intraoperative
  A "miss" is any alteration in surgical plan after review of FGC data to prevent decr sensitivity for the sentinel node (SN), or incr morbidity. Any change to surgical plan that results in a change of anatomic or incision location, or addition of lymph node (LN) location will qualify as a miss. Removal of "hot" LN based on MGC data that would not have been removed based on FGC imaging will not be counted as a "miss," incl non-localization of a SN by FGC imaging, provided they are within 10% of the counts of the "hottest" node.
Quantification of the time required to use the MGC imaging system for initial lymphoscintigraphy imaging | In minutes and seconds
The rate of agreement of hot spot detection between the FGC and MGC imaging systems. | intraoperative
  Recorded as a percentage of total hotspots detected between both modalities
Success rate of MGC imaging and the gamma probe in identifying SLNs independent of investigator review of FGC imaging findings | Intraoperative
  This is defined as the percentage of cases where the sentinel node was detected by the MGC and gamma probe surveys correctly prior to un-blinding to FGC images.
The number of cases where the MGC identifies a false negative, a false positive, clarifies ambiguous FGC imaging or provides other specific clinical advantages for completion of SLNBx | Intraoperative
  Descriptive statistics will be used to describe individual cases where the MGC provided information that would alter surgical decision making.

SECONDARY OUTCOMES:
Logistical issues of use of MGC imaging as currently configured. | Intraoperative and perioperative
  This is recorded on Likert score based surveys administered to the study surgeon regarding the logistic ease of the process of using the MGC devices.
Time required for standard FGC imaging and time required for MGC imaging in the preoperative suite (time data from the Department of Radiology will be used to calculate the average imaging time associated with FGC imaging). | Intraoperative and perioperative
Investigator identification of clinical scenarios where the hand-held gamma probe provided additional benefit to the MGC for pre-operative evaluation of hot spots. | Intraoperative
  Descriptive statistics will again be used to define specific cases where this occurred.
Ergonomic optimization of our method for intraoperative gamma imaging as measured by operative time and surgeon satisfaction. | Preoperative and intraoperative
  This will include specific changes to the MGC systems implemented to increase ease of use and sensitivity of the system.

CONTACTS AND LOCATIONS:
Overall Officials: Craig L Slingluff, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

REFERENCES:
- [Derived] Judge JM, Popovic K, Petroni GR, Kross B, McKisson J, McKisson J, Weisenberger AG, Stolin A, Majewski S, Rehm P, Slingluff CL, Williams MB, Dengel LT. Evaluation of Preoperative and Intraoperative Mobile Gamma Camera Imaging in Sentinel Lymph Node Biopsy for Melanoma Independent of Preoperative Lymphoscintigraphy. J Surg Res. 2023 May;285:176-186. doi: 10.1016/j.jss.2022.12.013. Epub 2023 Jan 20. PMID 36682343